CLINICAL TRIAL: NCT00039884
Title: Phase II Study of NESP (Novel Erythropoiesis Stimulating Protein) During Concurrent Chemo-Radiation for the Treatment of Cervical Carcinoma.
Brief Title: Will Radiation/Chemotherapy Treatment of Cervical Cancer Work Better With Medication That May Improve Anemia?
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mirhashemi, Ramin, M.D. (Individual)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 01/155A
Record Dates: First submitted 2002-06-13; First posted 2002-06-17 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-06

CONDITIONS: Anemia; Cervix Neoplasms
Keywords: Cervical cancer
MeSH Terms: conditions — Anemia; Uterine Cervical Neoplasms | interventions — Darbepoetin alfa

INTERVENTIONS:
Drug: NESP - Novel Erythropoiesis Stimulating Protein

SUMMARY:
This is a clinical trial (a type of research study) designed to describe the efficacy (effectiveness) and toxicity (safety) of a new medical treatment, NESP (Novel Erythropoiesis Stimulating Protein). This study will be offered to patients with cervical cancer undergoing a combination of chemotherapy and radiation. This treatment may lower your red blood cells. The use of NESP may stimulate the body to produce more red blood cells. Our hypothesis is that higher red blood cells will be beneficial to the patient during treatment for cervical cancer.

ELIGIBILITY:
* Consent form completed and signed
* Hemoglobin between 9-13 g/dL
* Life expectancy of at least 4 months
* Karnofsky Performance Status =/> 70
* No evidence of hemolysis, GI bleeding, or bleeding due to recent surgery
* Adequate renal and liver function

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64
Dates: Start 2001-09; Study Completion 2003-03

CONTACTS AND LOCATIONS:
Locations (1):
- Sylvester Comprehensive Cancer Center/JMH, Miami, Florida, United States